CLINICAL TRIAL: NCT04474860
Title: Study on Gene Mutation Spectrum of Malignant Hyperthermia in China Based on the Establishment of Bioinformatics Database
Brief Title: Gene Mutation Spectrum of Malignant Hyperthermia in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Bin Liu, Professor, West China Hospital
Other Study IDs: 2018HXFH006
Record Dates: First submitted 2020-07-13; First posted 2020-07-17 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Malignant Hyperthermia
Keywords: Malignant Hyperthermia; Gene mutation spectrum; Bioinformatics database
MeSH Terms: conditions — Malignant Hyperthermia | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Malignant Hyperthermia: Samples from Chinese whose malignant hyperthermia susceptibility had been confirmed after a positive clinical manifestation of malignant hyperthermia and samples from their blood relations will receive genetic testing.
  Interventions: Diagnostic Test: gene sequencing

INTERVENTIONS:
Diagnostic Test: gene sequencing — Gene fragment analysis, Sanger sequencing method and/or high-throughput whole-genome sequencing will be performed to find the pathogenic gene and mutation site of MH in Chinese population.

SUMMARY:
In this study, case information and specimens of patients with malignant hyperthermia(MH) will be collected from all over China, and gene fragment analysis, sanger sequencing method and/or high-throughput whole-genome sequencing will be performed. The MH bioinformatics database will be established to find the pathogenic gene and mutation site of MH in Chinese. Based on the bioinformatics database, the genetic law of MH family will be studied. According to the results of the study, the guideline for the diagnosis and treatment of MH that is in line with Chinese population biology characteristics will be formulated.

DETAILED DESCRIPTION:
When MH cases or suspected cases occur in China, anesthesiologists can seek help through malignant hyperthermia emergency rescue WeChat group in which experts from all over the country will give therapy instructions. Afterwards, the responsible anesthesiologist will complete the case report form (CRF) and collect family history of MH. The quality of CRF is reviewed by the investigator and all the queries are solved within 1~2 weeks.

Upon obtaining the informed consent, all biological specimens of MH confirmed or suspected patients and their blood relations will be collected in the local hospitals and transported to West China Hospital, Sichuan University in dry ice packaging. All specimens will be checked by the trained investigator, registered and labeled in a standardized manner, and then stored in the biological sample bank of West China Hospital, Sichuan University.

Firstly, investigators will use the method of gene fragment analysis to detect the samples at the diagnostic mutation sites included in the current European malignant hyperthermia group. Secondly, investigators will use sanger sequencing method to verify the mutation variants. If the screening results are negative, then high-throughput whole-genome sequencing will be performed.

The MH bioinformatics database will be established to find the pathogenic gene and mutation site of MH in Chinese. Based on the bioinformatics database, the genetic law of MH family will be studied. According to the results of the study, the guideline for the diagnosis and treatment of MH that is in line with Chinese population biology characteristics will be formulated.

ELIGIBILITY:
Inclusion Criteria:

* Chinese whose malignant hyperthermia susceptibility had been confirmed after a positive clinical manifestation of malignant hyperthermia which defined as their scores of clinical grading scale for malignant hyperthermia are more than 35 and their blood relations.
* Sign informed consent

Exclusion Criteria:

* Patients who have no adverse anaesthetic event, such as those patients referred with a history of exertional heat illness, exertional or recurrent rhabdomyolysis, or a congenital myopathy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clinically diagnosed MH patients in China and their blood relations
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Pathogenic gene and mutation site of MH in Chinese | Within data collection period (5 years total)
  Samples from patients with MH and their blood relations in China will be detected by gene fragment analysis and then verified by Sanger sequencing method and/or detected by high-throughput whole-genome sequencing to find the pathogenic gene and mutation site of MH in Chinese.

SECONDARY OUTCOMES:
Clinical profiles and outcomes of patients with MH in China | Within data collection period (5 years total)
  This study will summarize the Clinical profiles of patients with MH in China by collecting and analyzing case information of patients with MH from all over China.
The genetic law of MH family | Within data collection period (5 years total)
  Collecting samples from the MH patients and their blood relations and undertaking gene fragment analysis, Sanger sequencing method and/or high-throughput whole-genome sequencing, family genitive tree for MH will be then drawn.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Liu, MD, Principal Investigator — West China Hospital; Yunxia Zuo, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided